CLINICAL TRIAL: NCT05908266
Title: Behavioural Study of Reaching Control in Healthy Volunteers and Volunteers With Parkinson Disease in Dynamical Context
Brief Title: Flexible Reaching Control in Parkinson Disease
Acronym: REACH-PD
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: REACH-PD
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD: Patients with Parkinson disease
  Interventions: Other: Reaching movements; Other: Disease Assessment
- Control: Healthy volunteers
  Interventions: Other: Reaching movements

INTERVENTIONS:
Other: Reaching movements — Participants will be instructed to perform reaching movements by moving the handle of a robotic arm mounted with a virtual reality display.
Other: Disease Assessment — Disease stage assessed by trained professionals
  Groups: PD

SUMMARY:
Current research and theories have highlighted that the parameters linked to movement planning, e.g. the decision to select a movement goal, and adaptation, e.g. the ability to update control dependent on a novel dynamical context, are update quickly and within an ongoing movement in the general population. In parallel, it has been suggested that the evaluation of movement costs is a function of the basal ganglia, and it is impaired in Parkinson disease (PD). Here the investigators want to test whether these mechanisms also alter the ability of patients to update control during an ongoing action. A positive result would confirm that movement-related costs and dynamical representations depend on the integrity of the basal ganglia, in contrast a negative result would indicate that the deficit in PD is more specifically related to movement initiation, which would invite one to reconsider the cause of bradykinesia in this population.

ELIGIBILITY:
Inclusion Criteria:

* Ability to perform the task (assessed during the experiment)

Exclusion Criteria:

* Inability to perform the task (motor) or to understand the task requirements (cognitive)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be based on two populations: on population of volunteers with Parkinson disease, and one population of age and sex matched healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Kinematics | Measured during the entire experiment (an average of 4.5 years)
  Position of the handle as a function of time. Units are millimetres
Surface Electromyogram | Measured during the entire experiment (an average of 4.5 years)
  Surface recordings of muscles activities from the main muscles involved in movement production. Units are volts
Applied forces | Measured during the entire experiment (an average of 4.5 years)
  Forces applied by participants on the robotic handle. Units are Newtons

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Crevecoeur, PhD, Study Director — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No